CLINICAL TRIAL: NCT05685511
Title: Behavioral Activation and Medication Optimization For Improving Perioperative Mental Health In Older Adults Undergoing Oncologic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202212097; 1P50MH122351 (NIH)
Record Dates: First submitted 2023-01-05; First posted 2023-01-17 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Older Adults; Anxiety; Depression; Major Surgical Resection of a Thoracic Malignancy; Major Surgical Resection of an Abdominal Malignancy
Keywords: behavioral activation; medication optimization; thoracic surgery; oncologic surgery; perioperative mental health
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Study staff responsible for administering ratings throughout the study are blinded. This blinding is kept throughout the study until data collection is complete. At the end of the follow-up, the study coordinator will complete a blinding question to try to guess the arm to which each participant was allocated. This will allow to determine whether the blinding procedures in the study were effective.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator): Patients will receive resources either by mail or email. The resources include options for exploring brain health, supporting sleep and mental health, and introducing community resources for older adults.
  Interventions: Other: Usual care resources
- Intervention Bundle (Behavioral Activation + Medication Optimization) (Experimental): * Behavioral activation (BA) will span across 3 months postoperatively & will begin pre-operatively, with sessions approximately every two weeks. After discharge, the behavioral intervention will continue for 10-12 sessions, or out to approximately 3 months postoperatively.
  * Medications will be reviewed & optimized by a team of interventionists including a psychiatrist, pharmacologist, & pharmacists. While the participant is in-hospital, the interventionist's role will include coordinating with the hospital team to ensure that medication changes that were introduced preoperatively are maintained in-house & that no new inappropriate medications are initiated. After discharge, & up to approximately 3 months postoperatively, the interventionist will ensure that medication changes are reconciled during transitions of care. The interventionists will ensure the agreed-upon changes are implemented, or an alternative course of action is justified.
  Interventions: Behavioral: Behavioral Activation; Other: Medication Optimization

INTERVENTIONS:
Behavioral: Behavioral Activation — The behavioral intervention will consist of behavioral activation (BA), the basic premise of which is to help people with mental health problems to engage in activities that are reinforcing or meaningful and guided by their personal values
  Arms: Intervention Bundle (Behavioral Activation + Medication Optimization)
Other: Medication Optimization — Medication optimization consists of a simple set of principles: reconcile patient's medications, identify the patient's likely need for, and interest in, a medication adjustment, make the adjustment, and assess the response to that adjustment.
  Arms: Intervention Bundle (Behavioral Activation + Medication Optimization)
Other: Usual care resources — List of resources that the patient can explore on their own
  Arms: Usual Care

SUMMARY:
Using a Hybrid Type 1 Effectiveness-Implementation randomized control trial (RCT) design, the investigators will test the effectiveness of a bundled behavioral activation and medication optimization in reducing symptoms of depression and anxiety in older adults undergoing oncologic surgery (compared with usual care), while examining implementation outcomes.

ELIGIBILITY:
Inclusion Criteria:

Pre-screening:

To be considered for participation, patients will be screened using PHQ-4 questionnaire. Scores >3 will indicate positive pre-screen (i.e. can be considered for participation and formal screening). Scores < 3 will indicate negative screen (i.e. patient not considered for formal screening due to low risk for anxiety or depression).

Screening:

* Adults age ≥60 years
* Scheduled major thoracic, breast, or abdominal surgery for suspected or confirmed malignancy
* PHQ-ADS (Patient Health Questionnaire Anxiety and Depression Scale) ≥10 indicating clinically significant depression or anxiety symptoms.

Exclusion Criteria:

* Barrier to communication (Unable to read, speak, and understand English)
* Severe cognitive impairment screened by the SBT (Short Blessed Test) >10
* Acutely suicidal
* Considered ineligible per the discretion of the oncologic surgeon or study PI
* Previous participation in this study or another CPMH study of the intervention bundle or its feasibility.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2023-03-10 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2024-07-12 (Actual)

PRIMARY OUTCOMES:
Change in depression as measured by the Patient Health Questionnaire Anxiety and Depression Scale (PHQ-ADS) | Baseline, 1-month follow-up, and 3-month follow-up
  * 9 item questionnaire with answers ranging from 0=not at all to 3=nearly every day.
  * Scores represent: 0-5=mild, 6-10=moderate, 11-15=moderately severe, and 16-20=severe depression.
Change in anxiety as measured by the Patient Health Questionnaire Anxiety and Depression Scale (PHQ-ADS) | Baseline, 1-month follow-up, and 3-month follow-up
  * 7 item questionnaire with answers ranging from 0=not at all to 3=nearly every day. Total score for the seven items ranges from 0 to 21.
  * Scores 0-5=mild anxiety, 6-10=moderate anxiety, 11-15=moderately severe anxiety, and 15-21=severe anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin D Kozower, M.D., MPH, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holzer KJ, Bartosiak KA, Calfee RP, Hammill CW, Haroutounian S, Kozower BD, Cordner TA, Lenard EM, Freedland KE, Tellor Pennington BR, Wolfe RC, Miller JP, Politi MC, Zhang Y, Yingling MD, Baumann AA, Kannampallil T, Schweiger JA, McKinnon SL, Avidan MS, Lenze EJ, Abraham J. Perioperative mental health intervention for depression and anxiety symptoms in older adults study protocol: design and methods for three linked randomised controlled trials. BMJ Open. 2024 Apr 3;14(4):e082656. doi: 10.1136/bmjopen-2023-082656. PMID 38569683
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

DOCUMENTS (2):
  • Statistical Analysis Plan (2025-05-31): https://cdn.clinicaltrials.gov/large-docs/11/NCT05685511/SAP_003.pdf
  • Informed Consent Form (2024-01-05): https://cdn.clinicaltrials.gov/large-docs/11/NCT05685511/ICF_001.pdf